CLINICAL TRIAL: NCT03632707
Title: Role of Magnetic Resonance Imaging in the Diagnosis of Posterior Medial Meniscal Root Tear of the Knee
Brief Title: Magnetic Resonance Imaging of Medial Meniscal Posterior Root Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AAQardash, Principle Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRIOMMPRT
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-01

CONDITIONS: Medial Meniscus, Posterior Horn Derangement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic resonance imaging of the knee (Other): Patients complain of painful knee with clinical suspicious of medial meniscus posterior root tear of the knee will be examined by all Magnetic Resonance Imaging sequences including sagittal, coronal and axial PD,T2 and PD-SPIR weighted images, and correlate the results with Knee Arthroscopy.while the suspected cases of meniscal extrusion will make MRI using the knee coil for varus stress Overloading simulating weight bearing.
  Interventions: Radiation: Magnetic Resonance Imaging of the knee; Procedure: Knee Arthroscopy

INTERVENTIONS:
Radiation: Magnetic Resonance Imaging of the knee — After clinical assessment, all the patients will examined by Magnetic Resonance Imaging to diagnose the medial meniscal posterior root tear,and the suspected cases of meniscal extrusion will make MRI using the knee coil for varus stress Overloading simulating weight bearing
Procedure: Knee Arthroscopy — Correlate all the magnetic resonance imaging results with the Knee Arthroscopy

SUMMARY:
The aim of this study is to evaluate and analyze the role of magnetic resonance imaging in the diagnosis of medial meniscal posterior root tears, including the normal variations in meniscal anatomy that may resemble a meniscal tear, and identifying the causes or nature of posterior medial meniscal root tear(degenerative versus traumatic) and correlate the results with the standard reference knee Arthroscopy.In addition to identifying and estimating the suspected cases of meniscal extrusion by making MRI with stress varus overloading simulating weight bearing.

DETAILED DESCRIPTION:
The knee joint is one of the most important joints in the human body responsible for weight-bearing and a group of complex movements during ordinary life activities and even in vigorous sports making it susceptible to different traumatic injuries.Knee pain is considered as one of the most common complaints of patients presenting to clinical practitioners.There are many structures within the knee which can cause pain. By far, one of the most common causes of knee pain is a meniscus tear.The meniscus is the most important cushion in the knee; It plays an important bio mechanical role in axial load distribution of the knees. If the meniscus is injured and the cushioning is lost, arthritis and pain can occur.Menisci can tear due to traumatic injury or degenerative wear, meniscal root tears are a type of meniscal tear in the knee where the tear extends to either the anterior or posterior meniscal root attachment to the central tibial plateau. They often tend to be radial tears extending into the root.The medial meniscal posterior root tear can occur especially in middle-aged or older patients who have a single event of posteromedial painful popping sensation during light activities.Magnetic resonance imaging is well established as the best imaging modality for evaluating a patient with suspected meniscal pathology, involving the medial meniscal posterior horn root.In recent years, posterior meniscal root tears have received increasing attention in both Arthroscopic and Magnetic resonance study. All sequences of Magnetic resonance imaging should be reviewed, but T2 weighted coronal sections should provide the best visualization of the posterior roots. The Magnetic resonance findings of a medial meniscal posterior radial root tear are shortening or absence of the root (ghost sign) on sagittal images and a vertical fluid cleft with truncation sign and features of meniscal extrusion on coronal images.

It is very important to avoid errors in diagnosing meniscal root tears. So interpreting Magnetic resonance examinations of the knee need to be aware of the attachments of the menisci and to understand the normal variations in meniscal anatomy that may resemble a meniscal tear.

Tears of the meniscal root are relatively uncommon, occurring in 2.2% - 9.8% of patients undergoing Magnetic resonance imaging of the knee.However, it is important that these tears be diagnosed as several complications of meniscal root tear, including meniscal extrusion, secondary osteoarthritis, and subchondral insufficiency fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex from more than 16 years, having acute or chronic painful knee associated with popping sounds are included in this study.

Exclusion Criteria:

* Patients who are contraindicated to Magnetic Resonance Imaging examination as those who have artificial cardiac pacemaker or metallic prosthesis not compatible with Magnetic Resonance Imaging or those with severe claustrophobia.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Patients complain of painful knee joint associated with popping sounds and clinically suspected of medial meniscal posterior root tear will examined by Magnetic Resonance Imaging | 6 months
  Correlation the results of Magnetic Resonance Imaging with gold standard knee Arthroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Nisreen A. Abbas, MD, Study Director — Assiut University
Locations (1):
- Ashgan Ali Abdo Qardash, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barile A, Conti L, Lanni G, Calvisi V, Masciocchi C. Evaluation of medial meniscus tears and meniscal stability: weight-bearing MRI vs arthroscopy. Eur J Radiol. 2013 Apr;82(4):633-9. doi: 10.1016/j.ejrad.2012.10.018. Epub 2012 Nov 28. PMID 23199751
- [Result] Park HJ, Kim SS, Lee SY, Choi YJ, Chung EC, Rho MH, Kwag HJ. Medial meniscal root tears and meniscal extrusion transverse length ratios on MRI. Br J Radiol. 2012 Nov;85(1019):e1032-7. doi: 10.1259/bjr/26261821. PMID 23091292
- [Result] Carreau JH, Sitton SE, Bollier M. Medial Meniscus Root Tear in the Middle Aged Patient: A Case Based Review. Iowa Orthop J. 2017;37:123-132. PMID 28852346
- [Result] Costa CR, Morrison WB, Carrino JA. Medial meniscus extrusion on knee MRI: is extent associated with severity of degeneration or type of tear? AJR Am J Roentgenol. 2004 Jul;183(1):17-23. doi: 10.2214/ajr.183.1.1830017. PMID 15208101